CLINICAL TRIAL: NCT00083850
Title: Genetics and Cardiovascular Reactivity in Young Twins
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1256; R21HL076723 (NIH)
Record Dates: First submitted 2004-06-02; First posted 2004-06-04 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To evaluate the effects of genetic variants in all of the nine adrenergic receptor subtype genes, alone or in combination, on cardiovascular reactivity and other quantitative cardiovascular traits in a population of 1048 healthy young twins.

DETAILED DESCRIPTION:
BACKGROUND:

Several studies have shown that cardiovascular reactivity (CVR) to acute laboratory stress is a stable and heritable trait and predictive of future blood pressure (BP) levels and essential hypertension (EH). The sympathetic nervous system (SNS) has a major role in BP regulation and adrenergic receptor subtypes mediate BP responses to acute challenges. As such, our hypothesis is that individual differences in CVR are partly determined by variation in genes encoding for adrenergic receptors mediating the sympathoadrenal response to stress. There is increasing evidence that this cardiovascular response is regulated by multiple adrenoceptor subtypes with structural homology. To date, nine homologous adrenergic receptor subtypes have been described. Only one study has found a gene-gene interaction upon CV disease incorporating two adrenergic receptor subtypes. Genetic variants in all the nine adrenergic receptor subtypes have never before been investigated in a single study as this study will do.

DESIGN NARRATIVE:

The study will evaluate the effects of genetic variants in all of the nine adrenergic receptor subtype genes, alone or in combination, on CVR and other quantitative cardiovascular traits in a population of 1048 healthy youth. Subjects are black and white twins that have already been comprehensively phenotyped as part of the Georgia Cardiovascular Twin Study (HL56622). Racial differences in adrenoceptor gene effects will receive special attention, because such differences may offer a partial explanation for the higher prevalence of essential hypertension (EH) in blacks. Primary measures are systolic BP at rest and in response to two behavioral stressors. Secondary measures are diastolic BP, cardiac output and total peripheral resistance (TPR) at rest and in response to the stressors, left ventricular mass (LVM), endothelium dependent arterial dilation to reactive hyperemia (EDAD), arterial stiffness and 24-hour ambulatory BP. This data set will be expanded through collection of buccal cell DNA from the parents of the twins, enabling performance of TDTs (transmission disequilibrium tests) and haplotype reconstruction and analyses. This candidate gene study in a large group of black and white twins including TDT and haplotype analyses provides an innovative approach to help identify individuals at particular risk for the development of EH and improve options for primary prevention as well as individualized therapy of EH (pharmacogenetics).

ELIGIBILITY:
No eligibility criteria

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2004-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanbin Dong — Augusta University